CLINICAL TRIAL: NCT06443021
Title: Investigation of the Influence of Variable Fill Volume, Dwell Duration and Dialysis Fluid Glucose Composition on Measured Ultrafiltration Volume (UFV) in Automated Peritoneal Dialysis (APD) Patients
Brief Title: Influence of Variable Inflow Volume, Dwell Duration and Glucose Concentration on Ultrafiltration Volume in APD Patients
Acronym: pPD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal decision
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: Winicker Norimed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PD-pPD-01-ESP
Record Dates: First submitted 2024-05-17; First posted 2024-06-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Renal Failure; Chronic Kidney Diseases
Keywords: Renal replacement therapy; Peritoneal dialysis; Automated peritoneal dialysis; PD cycler
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Prospective, multi-centric, interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peritoneal dialysis (PD) (Other): During the clinical phase, patients are treated continuously with the PD cycler sleep•safe harmony.
  The total duration of the clinical for the individual patient comprises a maximum of 17 weeks starting from V0
  Interventions: Device: PD cycler

INTERVENTIONS:
Device: PD cycler — After a training phase and a run-in period of up to 6 weeks, depending on the PD cycler used prior to the study, the interventional phase will be initiated.
  * Study phase A, variation of dwell duration: Duration of short cycles (cycle 1 and 2) 30 min, 60 min, 90 min, 120 min (and 150 min depending on the patient´s constitution and at the discretion of the treating physician)
  * Study phase B, variation of dialysis fluid glucose composition: 1st cycle: 1.5% glucose concentration, 2nd cycle: 2.3% glucose concentration, 3rd cycle: 1.5% glucose concentration, 4th cycle: 2.3% glucose concentration; all following cycles to be applied as prescribed by the treating physician.
  * Study phase C, variation of fill volume: 60% fill volume, 80% fill volume, 100% fill volume and 120% fill volume. (Volume of 120% will only be applied in case the patient tolerates these volumes according to the IPP.

SUMMARY:
The purpose of the current investigation is to provide proof of concept for a future approach to improve UF prediction accuracy. While building on the ideas of the past, the concept is augmented by leveraging additional diagnostic technologies and digital data analytics methodologies.

DETAILED DESCRIPTION:
The primary objective of this study is:

- UFV determined per defined dwells with variable dwell duration, dialysis fluid glucose composition and inflow volumes

The secondary objectives of this study are:

* Mean daily UFV
* Defined laboratory parameter like urea, creatinine, glucose, sodium determined in blood and dialysate during the extended PET (in dialysate additionally determination: phosphate, albumin removal)
* Treatment parameter: performed treatment duration and volume
* Fluid status measured by Body Composition Monitor (BCM)
* Manual IPP determination during the extended PET: At the first half of the dwell (during the first hour) for every 20 min and during the second half after 2h, 3h and 4h dwell time
* Residual renal function (RRF): renal urea and creatinine clearance, 24h urine output, Glomerular filtration rate (GFR)
* Extended PET
* 24 h batch collection (including e.g. total peritoneal clearance)
* Analysis of daily dietetic fluid intake, weight and further parameters documented by the patient in a patient diary

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated by study patient and investigator/ authorized physician
* Patients between 18-65 of age
* Chronic kidney disease (CKD) patients being treated with nocturnal APD for at least 3 months
* Ability to understand the nature and requirements of the study
* Total Kt/V ≥ 1.7 (counting from recruitment of the patient the measurement should not be older than 3 months)
* APD patients using sleep•safe PD-cycler or sleep•safe harmony PD-cycler with an IPP ≤ 18 cm H2O for the fill volume of 120%

Exclusion Criteria:

* Any condition which could interfere with the patient's ability to comply with the study
* Patients who have any condition prohibiting the use of BCM, like patients with major amputations (e.g. lower leg)
* Patients who have been subject to peritonitis/ exit site infection during the last 4 weeks
* Women of childbearing age without effective means of contraception, pregnancy (pregnancy test will be conducted at start and end of study) or lactation period
* Life expectancy < 3 months
* Patients suffering from uncontrolled/ not well adjustable diabetes
* Recent history of drain related problems, catheter malfunction, or frequent alarms during treatment
* Patients with uncontrolled hypertension and/ or previous history of vascular instability during PD
* Patients treated with intermittent APD
* Participation in an interventional clinical study during the preceding 30 days
* Previous participation in the same study
* APD patients having dwell exchanges throughout the day ("day dwell")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Ultrafiltration volume (UFV) | every day during the 11 weeks treatment
  UFV determined per defined dwells with variable dwell duration, dialysis fluid glucose composition and inflow volumes.

SECONDARY OUTCOMES:
Fluid status | At study start, and then after 3 weeks, 4 weeks and 5 weeks.
  Fluid status measured by Body Composition Monitor (BCM)
24 h batch collection | At study start, and then after 3 weeks, 4 weeks and 5 weeks.
  RRF (24 h urine output)
24 h batch collection | At study start, and then after 3 weeks, 4 weeks and 5 weeks.
  RRF (GFR)
24 h batch collection | At study start, and then after 3 weeks, 4 weeks and 5 weeks.
  RRF (renal creatinine clearance)
24 h batch collection | At study start, and then after 3 weeks, 4 weeks and 5 weeks.
  RRF (renal urea clearance)
24 h batch collection | At study start, and then after 3 weeks, 4 weeks and 5 weeks.
  Peritoneal urea clearance
24 h batch collection | At study start, and then after 3 weeks, 4 weeks and 5 weeks.
  Peritoneal creatinine clearance

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Garcia Méndez, Dr., Principal Investigator — Hospital Son Espases

IPD SHARING:
Plan to Share IPD: No